CLINICAL TRIAL: NCT04847206
Title: Effects of MDMA-like Substances in Healthy Subjects
Acronym: MDMA-like
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2021-00405
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; 3,4-Methylenedioxyamphetamine; N(epsilon)-(malondialdehyde)lysine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 5-period cross-over design with four active substance conditions (equimolar doses of psychoactive substance) and placebo:
  1. MDMA (100 mg MDMA-hydrochloride; 84.1 mg MDMA free base) 2) MDA (93.9 mg MDA-hydrochloride; 78.0 mg MDA free base) 3) lysMDMA (171.7mg lysMDMA dihydrochloride; 84.1 mg MDMA free base) 4) lysMDA (165.6 mg lysMDA dihydrochloride; 78.0 mg MDA free base) 5) Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MDMA (100 mg MDMA-hydrochloride) (Experimental): MDMA (100 mg MDMA-hydrochloride; 84.1 mg MDMA free base)
  Interventions: Drug: 3,4-methylenedioxymethamphetamine
- MDA (93.9 mg MDA-hydrochloride) (Experimental): MDA (93.9 mg MDA-hydrochloride; 78.0 mg MDA free base)
  Interventions: Drug: 3,4-methylenedioxyamphetamine
- lysine-MDMA (171.7mg lysMDMA dihydrochloride (Experimental): lysine-MDMA (171.7mg lysMDMA dihydrochloride; 84.1 mg MDMA free base)
  Interventions: Drug: lysine-3,4-methylenedioxymethamphetamine
- lysine-MDA (165.6 mg lysMDA dihydrochloride; (Experimental): lysine-MDA (165.6 mg lysMDA dihydrochloride; 78.0 mg MDA free base)
  Interventions: Drug: lysine-3,4-methylenedioxyamphetamine
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine — A moderate dose of 100 mg MDMA will be administered.
  Other Names: MDMA
  Arms: MDMA (100 mg MDMA-hydrochloride)
Drug: 3,4-methylenedioxyamphetamine — A moderate dose of 93.9 mg MDA will be administered.
  Other Names: MDA
  Arms: MDA (93.9 mg MDA-hydrochloride)
Drug: lysine-3,4-methylenedioxymethamphetamine — A moderate dose of 171.7 mg lysine-MDMA will be administered.
  Other Names: lysine-MDMA
  Arms: lysine-MDMA (171.7mg lysMDMA dihydrochloride
Drug: lysine-3,4-methylenedioxyamphetamine — A moderate dose of 165.6 mg lysine-MDA will be administered.
  Other Names: lysine-MDA
  Arms: lysine-MDA (165.6 mg lysMDA dihydrochloride;
Other: Placebo — Placebo (Mannitol)
  Arms: Placebo

SUMMARY:
The serotonin (5-HT) and oxytocin releaser and so-called "empathogen" 3,4-methylenedioxymethamphetamine (MDMA) acutely produces positive feelings, empathy, and trust. MDMA is used recreationally (ecstasy), as research tool to study 5-HT and oxytocin function, and is investigated for MDMA-assisted psychotherapy.

MDMA is metabolized in part (10%) to the psychoactive metabolite 3,4-methylenedioxyamphetamine (MDA) which itself is also a recreational substance and has also been used to assist psychotherapy in the past. The present study aims to describe and directly compare for the first time the effects of MDMA and MDA in the same healthy volunteers and using modern psychological and psychometric tests.

Additionally, although amphetamines including MDMA and MDA induce mainly positive subjective effects they may also produce negative subjective drug effects including anxiety in particular at the onset of the subjective response and the rapid onset of euphoria may increase the risk of abuse. Additionally, blood pressure may increase rapidly at drug onset. A possible solution to mitigate anxiety, abuse-related rapid euphoria increases and/or rapid blood pressure changes at onset consist of slowing the onset of the drug effect by using a slow-release formulation of MDMA. In the present study, the investigators will characterize the effects of lysine-MDMA and lysine-MDA and compare their effects with MDMA/MDA to test the concept of attenuated effects across both substances.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA) is used as recreational substance (Ecstasy), research tool to stimulate serotonin (5-HT) and oxytocin release and study associated mood states, and as a potential therapeutic substance to enhance psychotherapy for post-traumatic stress disorder. MDMA is an amphetamine derivative which, unlike prototypical amphetamines, predominantly enhances serotonergic neurotransmission via release of 5-HT through the SERT and it less potently also releases dopamine and norepinephrine through the DA transporter and NE transporter, respectively. Furthermore, MDMA is known to trigger oxytocin release which may contribute to its effects to increase trust, prosociality, and enhance empathy. MDMA is therefore referred to as an "entactogen" or "empathogen". MDMA is currently the only empathogen investigated in substance-assisted psychotherapy but other substances including the MDMA-metabolite 3,4-methylenedioxyamphetamine (MDA) have been used in the past or may be used in the future.

Aim 1: MDA may exert greater perceptual psychedelic-like effects due to a more potent binding to the serotonin 5-HT2A receptor, and it may also act longer than MDMA partly due to a longer plasma half-life. However, effects of MDMA and MDA have never been compared directly in the same study in humans and there is only one modern study that characterized MDA in humans. Therefore, the present study aims to describe and directly compare for the first time the effects of MDMA and MDA in the same healthy volunteers using modern and sensitive psychological and psychometric tests.

Aim 2: Additionally, although amphetamines including MDMA and MDA induce mainly positive subjective effects they may also produce negative subjective drug effects including anxiety in particular at the onset of the subjective response and the rapid onset of euphoria may increase abuse liability. Additionally, blood pressure may increase rapidly at drug onset. A possible solution to mitigate anxiety, abuse-related rapid euphoria increases and/or rapid blood pressure changes at onset consist of slowing the onset of the drug effect by using a slow-release formulation of MDMA/MDA. Alternatively, amphetamines can be linked to the endogenous amino acid lysine forming inactive lysine-amphetamine which then liberates the active amphetamine slowly in the circulation via plasma peptidases. This approach has been implemented with the medication Lisdexamfetamine, which combines lysine with d-amphetamine. In the present study, the investigators will similarly characterize the effects of lysine-MDMA and lysine-MDA to test for attenuated effects across both substances in comparison with MDMA/MDA.

Using a two-factorial study design with four active substance conditions (MDMA vs. MDA and lysine-MDMA vs. lysine-MDA) the investigators will be able to test differences between MDMA and MDA (with and without lysine) as well as between lysinated a non-lysinated substance (regardless of active substance) in the same study and with high statistical power and within one study addressing two aims.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions to the end of the study days
7. Willing not to operate heavy machinery within 48 hours after substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance or MDMA use more than 20 times or use of any illicit substance within the previous two months (not including cannabis)
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Acute subjective effects I | 18 months
  Visual Analog Scales (VAS) assessing the intensity and duration of subjective effects on a scale from 0 - 100 percent with higher scores representing more intense effects
Plasma levels of MDMA | 18 months
  Assessed 18 times on each study day via blood samples
Plasma levels of MDA | 18 months
  Assessed 18 times on each study day via blood samples

SECONDARY OUTCOMES:
Acute Subjective effects II | 18 months
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely"
Acute Subjective effects III | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects
States of Consciousness Questionnaire | 18 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Psychological Insight Questionnaire | 18 months
  Assesses the degree of psychological insight caused by a psychedelic experience through 14-items to be answered on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Autonomic effects I | 18 months
  Assessed 20 times on each study day via systolic and diastolic blood pressure
Autonomic effects II | 18 months
  Assessed 20 times on each study day via heart rate
Autonomic effects III | 18 months
  Assessed 20 times on each study day via tympanic body temperature
Autonomic effects IV | 18 months
  Assessed 7 times on each study day via pupil diameter
Autonomic effects V | 18 months
  Assessed one time on each study day via ECG (QT-time)
Plasma levels of oxytocin | 18 months
  Assessed 5 times on each study day via blood samples
Emotion processing I | 18 months
  Assessed one time on each study day via Face Emotion Recognition Task (FERT).
Emotion processing II | 18 months
  Assessed one time on each study day via Multifaceted Empathy Test (MET).
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Freiburger Personality Inventory (FPI-R) | Baseline
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
HEXACO personality inventory | Baseline
  The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience. The HEXACO uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Defense Style Questionnaire (DSQ-40) | Baseline
  The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Straumann I, Vizeli P, Avedisian I, Erne L, Noorshams D, Vukalovic I, Eckert A, Luethi D, Rudin D, Liechti ME. Acute effects of MDMA, MDA, lysine-MDMA, and lysine-MDA in a randomized, double-blind, placebo-controlled, crossover trial in healthy participants. Neuropsychopharmacology. 2026 Jan;51(2):476-485. doi: 10.1038/s41386-025-02248-3. Epub 2025 Sep 25. PMID 40999236